CLINICAL TRIAL: NCT01679678
Title: A Double Blind, Randomized, Controlled Study, Performed in Subjects With Post Traumatic-post Surgical, Venus Insufficiency and Diabetic Hard to Heal/Chronic Wounds, to Evaluate the Safety and Efficacy of Polyheal-2 vs PolyHeal in Once Daily Regimen
Brief Title: A Study, Performed in Subjects With Post Traumatic-post Surgical ,Venus Insufficiency and Diabetic Hard to Heal/Chronic Wounds, to Evaluate the Safety and Efficacy of PolyHeal-2 Versus PolyHeal in Once Daily Regimen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business considerations
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MWPH-2012-08-01
Record Dates: First submitted 2012-08-20; First posted 2012-09-06 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Surgical Wound Dehiscence
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PolyHeal 2 (Experimental): Negatively charged 5-micron polystyrene microspheres in Water For Injection
  Interventions: Device: PolyHeal 2
- PolyHeal (Active Comparator): Negatively charged 5-micron polystyrene microspheres suspended in Dulbecco's Modified Eagle's Medium (DMEM)
  Interventions: Device: Polyheal

INTERVENTIONS:
Device: PolyHeal 2 — PolyHeal is a sterile medical device
  Other Names: PolyHeal; PolyHeal is a sterile medical device
  Arms: PolyHeal 2
Device: Polyheal — PolyHeal is a sterile medical device that is comprised of negatively charged 5-micron polystyrene microspheres suspended in
  Other Names: PolyHeal is a sterile medical device that is comprised of negatively charged 5-micron polystyrene microspheres suspended in DMEM
  Arms: PolyHeal

SUMMARY:
This is a double-blind , randomized, controlled, two-arm study aiming to evaluate the safety and efficacy of Polyheal-2 vs PolyHeal, in once daily application as compared to historical control. The study will enroll adult subjects with post traumatic/post surgical, venus insufficiency and diabetic hard to heal wounds who meet the entrance criteria which will be followed for 12 weeks.

DETAILED DESCRIPTION:
Subjects will undergo screenibg period of up to two weeks. Following to eligibilidy confirmation subjects will be randomized into one of the two treatment groups and treated with study device once daily for 4 weeks.

Continuation of study device for additional period is based on wound healing progression and under investigator's discretion.

Subjects will be followed up weekly following to 4 weeks of active treatment for additional 8 weeks untol week 12.

ELIGIBILITY:
Inclusion Criteria:

* Hard to heal/chronic post traumatic post surgical ,venus insufficiency and diabetic wound refractory to healing at least 4 weeks prior to study treatment (one or more target wound/s will be eligible per each subject to be treated by the same agent)
* Subjects who are able to read, understand, and sign the informed consent form. In case of compromised mental capacity, approval and signature of a legal guardian is required.

Exclusion Criteria:

* Presence of a systemic infection or significant local infection with copious purulent drainage, fluids drainage, gangrene, or cellulites, or necrosis at the target wound site, as well as nonviable tissue, sinus tracts or tunnels that cannot be removed by debridement.
* Wounds with exposed bones, tendons or ligaments
* Wounds with exposed orthopedic implants
* Wounds with exposed breast prostheses
* Uncontrolled diabetes with HbA1c >11%
* Subjects with BMI greater than 35kg/m2
* Woman who are pregnant or nursing, or of childbearing potential and are not using adequate contraception
* Participation in another clinical drug/device trial within 30 days prior to the Screening visit or during this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Achievement of at least (≥)75% viable granulation tissue (grade 7 or 8 on the granulometer scale) after 4 weeks of study treatment (active phase) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alex Berezovsky, MD, Principal Investigator — Head of Department of Plastic and reconstructive surgery; Eyal Gur, MD, Principal Investigator — Head of Plastic and Reconstructive Surgery Department, Souraski Medical Center; Leonid Kogan, MD, Principal Investigator — Head of Plastic Surgery Department Western Galilee Hospital; Yehuda Ulman, Proffesor, Principal Investigator — Head of Plastic surgery department ,Rambam Medical Center
Locations (4):
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Western Galilee Hospital, Nahariya
  - Souraski Medical Center, Tel Aviv